CLINICAL TRIAL: NCT02278328
Title: Magnetoencephalography / Magnetic Resonance Spectroscopy Dose Response Study of Arbaclofen in Autism Spectrum Disorder
Brief Title: MEG Study of Acute STX209 Effects in ASD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Timothy Roberts (Other)
Collaborators: Simons Foundation (Other); Clinical Research Associates, LLC (Other)
Responsible Party: Sponsor-Investigator, Timothy Roberts, Oberkircher Family Chair in Pediatric Radiology Vice-Chair Radiology Research Children's Hospital of Philadelphia, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 14-010857
Record Dates: First submitted 2014-10-17; First posted 2014-10-30 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-09

CONDITIONS: Autism Disorder
Keywords: dose titration study; electrophysiology
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Intervention Model Description: All subjects receive placebo and two separate doses of STX209 (15mg, 30mg). The order of administration of these (at weekly intervals) is randomized into groups: (A) placebo, 15, 30 ; (B) 15, placebo, 30 and (C) 15, 30, placebo.
Masking Description: Each participant receives dose of drug or placebo. Both participant and investigator are masked to dose level/placebo. It is not open label.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A. Placebo then 15mg then 30mg (Experimental): Subjects will receive a single dose of placebo on week 1, 15 mg of STX209 on week 2 and 30 mg of STX209 on week 3.
  Subjects will receive STX209 via oral disintegrating tablets, administered in individual 15mg tablets.
  Interventions: Drug: STX209 (15mg); Drug: placebo; Drug: STX209 (30mg)
- B. 15mg then placebo then 30mg (Experimental): Subjects will receive a single dose of 15 mg of STX209 on week 1, placebo on week 2 and 30 mg of STX209 on week 3.
  Subjects will receive STX209 via oral disintegrating tablets, administered in individual 15mg tablets.
  Interventions: Drug: STX209 (15mg); Drug: placebo; Drug: STX209 (30mg)
- C. 15mg then 30mg then placebo (Experimental): Subjects will receive a single dose of 15 mg of STX209 on week 1, 30 mg of STX209 on week 2 and placebo on week 3.
  Subjects will receive STX209 via oral disintegrating tablets, administered in individual 15mg tablets.
  Interventions: Drug: STX209 (15mg); Drug: placebo; Drug: STX209 (30mg)

INTERVENTIONS:
Drug: STX209 (15mg) — A randomized acute dose-response design will be employed with a total study duration of 3 weeks. At each visit, baseline MEG will be obtained followed by acute single-dose drug/placebo administration, followed 60 minutes later by repeat MEG. Each participant will receive a single dose of placebo in random order and a single dose of STX209 from smallest to largest (15mg, and 30mg). MRI and MRS will be performed immediately following MEG to provide an anatomic basis for source localization as well as to assess acute effects of STX209 administration on MRS estimates of GABA and glutamate. The STX209 (15mg) intervention is the "low dose"
  Other Names: Arbaclofen (15mg)
Drug: placebo — A randomized acute dose-response design will be employed with a total study duration of 3 weeks. At each visit, baseline MEG will be obtained followed by acute single-dose drug/placebo administration, followed 60 minutes later by repeat MEG. Each participant will receive a single dose of placebo in random order and a single dose of STX209 from smallest to largest (15mg, and 30mg). MRI and MRS will be performed immediately following MEG to provide an anatomic basis for source localization as well as to assess acute effects of STX209 administration on MRS estimates of GABA and glutamate. The placebo intervention is the non-active placebo control dose
Drug: STX209 (30mg) — A randomized acute dose-response design will be employed with a total study duration of 3 weeks. At each visit, baseline MEG will be obtained followed by acute single-dose drug/placebo administration, followed 60 minutes later by repeat MEG. Each participant will receive a single dose of placebo in random order and a single dose of STX209 from smallest to largest (15mg, and 30mg). MRI and MRS will be performed immediately following MEG to provide an anatomic basis for source localization as well as to assess acute effects of STX209 administration on MRS estimates of GABA and glutamate. The STX209 (30mg) intervention is the "high dose"
  Other Names: Arbaclofen (30mg)

SUMMARY:
This is a single-site, randomized, acute dose-response study to determine whether STX209 produces a dose-dependent significant change in MEG target parameters compared to baseline as well as compared to placebo treatment.

DETAILED DESCRIPTION:
Recent evidence from magnetoencephalographic (MEG) studies in ASD have pointed to abnormalities (specifically, delays) in auditory evoked neuromagnetic responses (e.g. M100 - see Roberts et al., 2010, and mismatch field, MMF - see Roberts et al., 2011) as well as abnormalities in the oscillatory behavior of auditory cortex, especially in the gamma band (30-50Hz), at rest and in response to simple auditory stimuli (see Gandal et al., 2010 and Cornew et al., 2012; Edgar et al., 2013). The local circuitry underlying such evoked activity and oscillations, and synaptic transmission in general, requires an appropriate balance of excitation and inhibition, mediated by glutamate and GABA, respectively. One model of the neural oscillatory deficits in ASD suggests that impaired regulatory control by inhibitory interneurons onto pyramidal cells underlies abnormal auditory latency and oscillatory electrophysiological measures. As such, electrophysiological deficits are interpreted in terms of local circuitry abnormalities, with inferences at the molecular level of imbalances in the activity of glutamate and GABA.

A candidate therapeutic for ASD has been developed - STX209, a GABA-B agonist. Since this pharmaceutical targets synaptic activity that has clear electrophysiological correlates, one goal of this proposal is to assess the responsiveness (sensitivity to change) of MEG measures to acute administration of STX209 at various doses in adolescents on the autism spectrum. The study also aims to establish the nature of the putative relationship between such electrophysiologic markers and GABA and glutamate levels using MEGAPRESS spectrally-edited magnetic resonance spectroscopy (MRS).

ELIGIBILITY:
Inclusion Criteria:

1. Right- handed males aged 14 to 17.75 years.
2. Diagnosis of ASD with the last 12 months according to the DSM-IV criteria, including Autistic Disorder, Pervasive Developmental Disorder - Not Otherwise Specified (PDD-NOS), and Asperger's Syndrome but excluding Childhood Dis-integrative Disorder and Rett Syndrome.
3. Current pharmacological treatment regimen has been stable for at least 4 weeks prior to Screening.
4. If the subject is already receiving stable non-pharmacological educational, behavioral, and/or dietary interventions, participation in these programs must have been continuous during the 2 months prior to Screening and subjects or their parent/caregiver may not electively initiate new or modify ongoing interventions for the duration of the study. Typical school vacations are not considered modifications of stable programming.
5. Prior to the conduct of any study-specific procedures, the subject must provide verbal assent to participate in the study (if developmentally appropriate), and the parent/caregiver must provide written informed consent. If the caregiver attending the clinic visits is not the parent, written consent must be obtained from the parent for the caregiver's participation in the study.

Exclusion Criteria:

1. No known neurological impairment (e.g., head trauma with loss of consciousness for more than 10 minutes, stroke, seizure disorder).
2. Claustrophobia
3. Metallic implanted prosthetic or stimulation device (including pacemaker)
4. Excessive metallic dental work (including braces, non-removable retainers)
5. Subjects who are currently receiving treatment with racemic baclofen, vigabatrin, tiagabine, or riluzole.
6. Subjects who have taken another investigational drug within the last 30 days.
7. Subjects who are not able to take oral medications.
8. Subjects who have a history of hypersensitivity to racemic baclofen.
9. Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Ages: 14 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2016-02; Primary Completion 2018-07-30 (Actual); Study Completion 2019-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Roberts, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Phladelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- A. Placebo Then 15mg Then 30mg: Subjects will receive a single dose of placebo, then (a week later) 15mg STX209 then (a week later) 30mg STX209. Subjects will receive STX209 via oral disintegrating tablets, administered in individual 15mg tablets.
  A randomized acute dose-response design will be employed with a total study duration of 3 weeks. At each visit, baseline MEG will be obtained followed by acute single-dose drug/placebo administration, followed 60 minutes later by repeat MEG. Over the course of the three weeks, each participant will receive a single dose of placebo and a single dose of STX209 from smallest to largest (15mg, and 30mg). On each occasion, separated by 1 week, participants will receive either placebo or 15mg STX209 or 30mg STX209. MRI and MRS will be performed immediately following MEG to provide an anatomic basis for source localization as well as to assess acute effects of STX209 administration on MRS estimates of GABA and glutamate.
- B. 15mg Then Placebo Then 30mg: Subjects will receive a single dose of 15mg STX209, then (a week later) placebo then (a week later) 30mg STX209. Subjects will receive STX209 via oral disintegrating tablets, administered in individual 15mg tablets.
  A randomized acute dose-response design will be employed with a total study duration of 3 weeks. At each visit, baseline MEG will be obtained followed by acute single-dose drug/placebo administration, followed 60 minutes later by repeat MEG. Over the course of the three weeks, each participant will receive a single dose of placebo and a single dose of STX209 from smallest to largest (15mg, and 30mg). On each occasion, separated by 1 week, participants will receive either placebo or 15mg STX209 or 30mg STX209. MRI and MRS will be performed immediately following MEG to provide an anatomic basis for source localization as well as to assess acute effects of STX209 administration on MRS estimates of GABA and glutamate.
- C. 15mg Then 30mg Then Placebo: Subjects will receive a single dose of 15mg STX209, then (a week later) 30mg STX209 then (a week later) placebo . Subjects will receive STX209 via oral disintegrating tablets, administered in individual 15mg tablets.
  A randomized acute dose-response design will be employed with a total study duration of 3 weeks. At each visit, baseline MEG will be obtained followed by acute single-dose drug/placebo administration, followed 60 minutes later by repeat MEG. Over the course of the three weeks, each participant will receive a single dose of placebo and a single dose of STX209 from smallest to largest (15mg, and 30mg). On each occasion, separated by 1 week, participants will receive either placebo or 15mg STX209 or 30mg STX209. MRI and MRS will be performed immediately following MEG to provide an anatomic basis for source localization as well as to assess acute effects of STX209 administration on MRS estimates of GABA and glutamate.
Period: Neuropsych Screening
Arm/Group | A. Placebo Then 15mg Then 30mg | B. 15mg Then Placebo Then 30mg | C. 15mg Then 30mg Then Placebo
Started | 10 | 7 | 8
Completed | 9 | 6 | 6
Not Completed | 1 | 1 | 2
Not completed — found ineligible on neuropsych | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — incomplete consent | 0 | 0 | 2
Period: First Intervention (1 Day)
Arm/Group | A. Placebo Then 15mg Then 30mg | B. 15mg Then Placebo Then 30mg | C. 15mg Then 30mg Then Placebo
Started | 9 | 6 | 6
Completed | 9 | 6 | 6
Not Completed | 0 | 0 | 0
Period: Washout (1 Week)
Arm/Group | A. Placebo Then 15mg Then 30mg | B. 15mg Then Placebo Then 30mg | C. 15mg Then 30mg Then Placebo
Started | 9 | 6 | 6
Completed | 9 | 6 | 6
Not Completed | 0 | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | A. Placebo Then 15mg Then 30mg | B. 15mg Then Placebo Then 30mg | C. 15mg Then 30mg Then Placebo
Started | 9 | 6 | 6
Completed | 9 | 6 | 6
Not Completed | 0 | 0 | 0
Period: Second Washout (1 Week)
Arm/Group | A. Placebo Then 15mg Then 30mg | B. 15mg Then Placebo Then 30mg | C. 15mg Then 30mg Then Placebo
Started | 9 | 6 | 6
Completed | 9 | 6 | 6
Not Completed | 0 | 0 | 0
Period: Third Intervention (1 Day)
Arm/Group | A. Placebo Then 15mg Then 30mg | B. 15mg Then Placebo Then 30mg | C. 15mg Then 30mg Then Placebo
Started | 9 | 6 | 6
Completed | 9 | 6 | 6
Not Completed | 0 | 0 | 0
Period: Third Washout (1 Week)
Arm/Group | A. Placebo Then 15mg Then 30mg | B. 15mg Then Placebo Then 30mg | C. 15mg Then 30mg Then Placebo
Started | 9 | 6 | 6
Completed | 9 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Subjects receive a single dose of STX209 or placebo starting at 15 mg, increasing to 30 mg on each of three separate occasions (different dose on each occasion, according to their randomization scheme Arm. Outcome measures are reported by dose administered (or placebo) and not by randomization schedule, since the same outcome measures are acquired after each dose administration. Subjects will receive STX209 via oral disintegrating tablets, administered in individual 15mg tablets.
  A randomized acute dose-response design is employed with a total study duration of 3 weeks. At each visit, baseline MEG will be obtained followed by acute single-dose drug/placebo administration, followed 60 minutes later by repeat MEG. MRI and MRS will be performed immediately following MEG to provide an anatomic basis for source localization as well as to assess acute effects of STX209 administration on MRS estimates of GABA and glutamate.
Arm/Group | All Participants
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.8 (.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 21
M50 Latency (Left Hemisphere) [Mean (Standard Deviation); unit: ms] — Latency of M50 evoked response component arising from left cerebral hemisphere Population: in 2 cases pre-placebo and in 1 case each pre-15mg and pre-30mg, evoked response data was unevaluable due to artifact
  ms
    Pre-placebo: number analyzed (Participants) | 19
    Pre-placebo | 89.9 (19.2)
    Pre-15mg dose: number analyzed (Participants) | 20
    Pre-15mg dose | 91.9 (15.0)
    Pre-30mg dose: number analyzed (Participants) | 20
    Pre-30mg dose | 90.8 (13.9)
M50 Latency (Right Hemisphere) [Mean (Standard Deviation); unit: ms] — Latency of M50 evoked response component arising from right cerebral hemisphere Population: in 2 cases pre-placebo,1 case pre-15mg and and 2 cases pre-30mg, evoked response data was unevaluable due to artifact
  ms
    Pre-placebo: number analyzed (Participants) | 19
    Pre-placebo | 95.6 (24.0)
    Pre-15mg dose: number analyzed (Participants) | 20
    Pre-15mg dose | 96.9 (27.6)
    Pre-30mg dose: number analyzed (Participants) | 19
    Pre-30mg dose | 93.6 (21.6)
Steady State Inter-Trial Coherence (Left Hemisphere) [Mean (Standard Deviation); unit: unitless] — inter-trial coherence (ITC) of left hemisphere responses to steady state auditory stimuli Population: in 1 participant prior to 15mg and in 4 participants prior to 30mg dose, data was unevaluable.
  unitless
    Pre-placebo | .214 (.122)
    Pre-15mg dose: number analyzed (Participants) | 20
    Pre-15mg dose | .237 (.106)
    Pre-30mg dose: number analyzed (Participants) | 17
    Pre-30mg dose | .239 (.129)
Steady State Inter-Trial Coherence (Right Hemisphere) [Mean (Standard Deviation); unit: unitless] — Inter-trial coherence (ITC) to auditory steady state stimuli arising from right cerebral hemisphere Population: in 1 participant prior to 15mg and in 4 participants prior to 30mg dose, data was unevaluable.
  unitless
    Pre-placebo | .273 (.168)
    Pre-15mg dose: number analyzed (Participants) | 20
    Pre-15mg dose | .316 (.181)
    Pre-30mg dose: number analyzed (Participants) | 17
    Pre-30mg dose | .321 (.173)
GABA (Left Hemisphere) [Mean (Standard Deviation); unit: ratio] — GABA/Cr ratio for voxel in left superior temporal gyrus Population: In 7 cases pre-placebo and in 5 cases each pre-15mg or 30mg, spectroscopy data was unevaluable
  ratio
    Pre-placebo: number analyzed (Participants) | 14
    Pre-placebo | .149 (.075)
    Pre-15mg dose: number analyzed (Participants) | 16
    Pre-15mg dose | .154 (.078)
    Pre-30mg dose: number analyzed (Participants) | 16
    Pre-30mg dose | .148 (.061)

OUTCOME MEASURES:

1. Primary Outcome: M50 Latency (Left Hemisphere)
Description: The latency of the M50 auditory evoked response component arising from the left cerebral hemisphere
Time Frame: 1 hour per intervention followed by a 1 week washout for a total of three weeks
Population: For placebo and 15mg dose, 1 case each was unavailable due to artifact. At 30mg dose, 2 cases were unevaluable due to artifact
Measure: Mean (Standard Deviation); unit: ms
Groups:
- All Participants: Results post placebo and each dose (15 and 30mg)
Arm/Group | All Participants
Number analyzed (Participants) | 21
ms
  Post placebo: number analyzed (Participants) | 20
  Post placebo | 90.9 (13.8)
  Post-15mg dose: number analyzed (Participants) | 20
  Post-15mg dose | 87.4 (16.9)
  Post-30mg dose: number analyzed (Participants) | 19
  Post-30mg dose | 89.3 (13.5)

2. Primary Outcome: M50 Latency (Right Hemisphere)
Description: The latency of the M50 auditory evoked response component arising from the right cerebral hemisphere
Time Frame: 1 hour per intervention followed by a 1 week washout for a total of three weeks
Population: For placebo and 15mg dose, 1 case each was unavailable due to artifact. At 30mg dose, 4 cases were unevaluable due to artifact
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | All Participants
Number analyzed (Participants) | 21
ms
  Post-placebo: number analyzed (Participants) | 20
  Post-placebo | 95.1 (21.7)
  Post-15mg dose: number analyzed (Participants) | 20
  Post-15mg dose | 87.8 (8.6)
  Post-30mg dose: number analyzed (Participants) | 17
  Post-30mg dose | 93.8 (23.6)

3. Primary Outcome: Steady State Inter Trial Coherence (Left Hemisphere)
Description: The inter trial coherence (ITC) of auditory steady state response arising from the left cerebral hemisphere
Time Frame: 1 hour per intervention followed by a 1 week washout for a total of three weeks
Population: For placebo, 3 cases and for 15mg and 30mg doses, 1 case each was unevaluable due to artifact.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | All Participants
Number analyzed (Participants) | 21
unitless
  Post-placebo: number analyzed (Participants) | 18
  Post-placebo | .253 (.134)
  Post-15mg dose: number analyzed (Participants) | 20
  Post-15mg dose | .239 (.111)
  Post-30mg dose: number analyzed (Participants) | 20
  Post-30mg dose | .244 (.116)

4. Primary Outcome: Steady State Inter Trial Coherence (Right Hemisphere)
Description: The inter trial coherence (ITC) of auditory steady state response arising from the right cerebral hemisphere
Time Frame: 1 hour per intervention followed by a 1 week washout for a total of three weeks
Population: For placebo, 3 cases and for 15mg dose and 30mg doses, 1 case each was unevaluable due to artifact.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | All Participants
Number analyzed (Participants) | 21
unitless
  Post-placebo: number analyzed (Participants) | 18
  Post-placebo | .324 (.178)
  Post-15mg dose: number analyzed (Participants) | 20
  Post-15mg dose | .325 (.166)
  Post-30mg dose: number analyzed (Participants) | 20
  Post-30mg dose | .306 (.153)

5. Primary Outcome: GABA (Left Hemisphere)
Description: GABA/Cr ratio arising from a voxel in the left superior temporal gyrus
Time Frame: 1 hour per intervention followed by a 1 week washout for a total of three weeks
Population: For placebo, 5 cases were unevaluable. For 15mg, 7 cases were unevaluable. For 30mg, 4 cases were unevaluable
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | All Participants
Number analyzed (Participants) | 21
ratio
  Post-placebo: number analyzed (Participants) | 16
  Post-placebo | .155 (.045)
  Post-15mg dose: number analyzed (Participants) | 14
  Post-15mg dose | .154 (.056)
  Post-30mg dose: number analyzed (Participants) | 17
  Post-30mg dose | .164 (.062)

ADVERSE EVENTS:
Time Frame: 3 weeks
Description: Although 25 participants are in the participant flow, two participants did not proceed past teh neuropsychological evaluation and onto any of the interventions and therefore did not receive any drug dose or placebo (having withdrawn or been excluded after screening). Therefore, we consider only 23 participants to have been placed at risk by the study.
Groups:
- Placebo: Subjects will receive a single dose of placebo via oral disintegrating tablets, administered as two individual tablets.
- STX209 (15mg): Subjects will receive a single dose of 15mg STX209 via oral disintegrating tablets, administered as two individual tablets (one being 15mg drug, one being placebo)
- STX209 (30mg): Subjects will receive a single dose of 15mg STX209 via oral disintegrating tablets, administered as two individual tablets (each being 15mg drug)
Arm/Group | Placebo | STX209 (15mg) | STX209 (30mg)
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 7/23 | 11/23 | 4/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=23) | STX209 (15mg) (N=23) | STX209 (30mg) (N=23)
cold symptoms / upper respiratory (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 1 (1) — stuffy nose, sore throat, coughing, sneezing
fatigue (General disorders) | 3 (3) | 4 (4) | 1 (1)
increased appetite (General disorders) | 1 (1) | 2 (2) | 0 (0) — hungry / thirsty
overly energetic (General disorders) | 2 (2) | 2 (2) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/28/NCT02278328/Prot_SAP_000.pdf